CLINICAL TRIAL: NCT06844058
Title: Efficacy of Islamic-Oriented Ericksonian Hypnotherapy vs. Standard Ericksonian Hypnotherapy in Reducing Anxiety and Depression: A Randomized Controlled Trial
Brief Title: Islamic-Oriented vs. Standard Ericksonian Hypnotherapy for Anxiety and Depression
Acronym: IEH-RTC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Nisantasi University (Other)
Responsible Party: Principal Investigator, Metin Çınaroğlu, Principal Investigator, Istanbul Nisantasi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IEH
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Anxiety Disorders; Depressive Disorder
Keywords: Hypnotherapy; Ericksonian Hypnosis; Islamic Psychology; Anxiety Reduction; Depression Treatment; Culturally Adapted Psychotherapy; Religious-Based Therapy
MeSH Terms: conditions — Anxiety Disorders; Depressive Disorder

STUDY DESIGN:
Intervention Model Description: This study follows a parallel-group randomized controlled design, where participants are assigned to one of three groups: Islamic-Oriented Ericksonian Hypnotherapy (IEH), Standard Ericksonian Hypnotherapy (SEH), or a control group with no intervention. Each participant remains in the same group throughout the study period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Islamic-Oriented Ericksonian Hypnotherapy (IEH) Group (Experimental): Participants receive 12 weekly sessions of Islamic-Oriented Ericksonian Hypnotherapy (IEH), which integrates faith-based imagery, Quranic metaphors, and religiously adapted hypnotic suggestions alongside standard Ericksonian techniques. Each session lasts 60 minutes.
  Interventions: Behavioral: Islamic-Oriented Ericksonian Hypnotherapy (IEH)
- Standard Ericksonian Hypnotherapy (SEH) Group (Active Comparator): Participants receive 12 weekly sessions of Standard Ericksonian Hypnotherapy (SEH), using metaphorical storytelling, indirect suggestions, guided imagery, and hypnotic language patterns without religious integration. Each session lasts 60 minutes.
  Interventions: Behavioral: Standard Ericksonian Hypnotherapy (SEH)
- Control Group (No Intervention) (No Intervention): Participants do not receive any intervention but will complete assessments at baseline, post-intervention (Week 12), and follow-up (Week 16).

INTERVENTIONS:
Behavioral: Islamic-Oriented Ericksonian Hypnotherapy (IEH) — This intervention involves 12 weekly sessions (60 minutes each) of Ericksonian hypnotherapy integrated with Islamic religious elements. Sessions incorporate:
  Quranic metaphors and Islamic imagery Spiritual affirmations to enhance relaxation and emotional regulation Faith-based guided hypnosis adapted to cultural and religious beliefs Techniques such as indirect suggestions, therapeutic storytelling, and guided imagery The intervention is designed for Muslim participants with mild to moderate anxiety and depression.
  Arms: Islamic-Oriented Ericksonian Hypnotherapy (IEH) Group
Behavioral: Standard Ericksonian Hypnotherapy (SEH) — Participants receive 12 weekly sessions (60 minutes each) of standard Ericksonian hypnotherapy, which includes:
  Metaphorical storytelling and guided imagery Indirect hypnotic suggestions to promote psychological flexibility Relaxation techniques to reduce anxiety and depressive symptoms Unlike the Islamic-Oriented Hypnotherapy (IEH), this intervention does not integrate religious or faith-based elements.
  Arms: Standard Ericksonian Hypnotherapy (SEH) Group

SUMMARY:
This randomized controlled trial (RCT) aims to compare the effectiveness of Islamic-Oriented Ericksonian Hypnotherapy (IEH) and Standard Ericksonian Hypnotherapy (SEH) in reducing symptoms of anxiety and depression. The study will enroll 90 participants with mild to moderate anxiety and depression, who will be randomly assigned to one of three groups: (1) IEH intervention, (2) SEH intervention, or (3) control group (no intervention). Participants in the intervention groups will receive 12 weekly hypnotherapy sessions, each lasting 60 minutes. The primary outcomes include changes in Beck Depression Inventory-II (BDI-II) and Beck Anxiety Inventory (BAI) scores from baseline to post-intervention and at a 4-week follow-up.

The study will also assess whether religious belief levels moderate the effects of the intervention using the OK-Religious Attitude Scale. Data collection will be performed at Istanbul Nişantaşı University, and ethical approval has been obtained.

DETAILED DESCRIPTION:
This randomized controlled trial evaluates the differential effects of Islamic-Oriented Ericksonian Hypnotherapy (IEH) and Standard Ericksonian Hypnotherapy (SEH) in alleviating symptoms of anxiety and depression among religious Muslim adults. The primary objective is to examine whether the integration of Islamic religious elements into Ericksonian hypnotherapy enhances clinical outcomes compared to its standard application.

The study follows a parallel-group design with three arms: IEH, SEH, and a no-intervention control. Ninety participants (30 per group) are randomized using stratified block randomization based on age and gender. All intervention sessions are manualized, delivered by trained clinical psychologists, and conducted weekly over 12 weeks (each lasting 60 minutes).

IEH sessions incorporate culturally and religiously adapted therapeutic elements, such as Quranic metaphors, Islamic imagery, and spiritual affirmations, in line with the Ericksonian framework. SEH sessions utilize traditional hypnotic techniques including metaphorical storytelling, guided imagery, and indirect suggestions, without religious content.

Primary outcome measures include changes in Beck Depression Inventory-II (BDI-II) and Beck Anxiety Inventory (BAI) scores from baseline to Week 12 (post-intervention) and Week 16 (follow-up). Secondary analyses will investigate whether religiosity levels (measured via the OK-Religious Attitude Scale) moderate treatment effects. Blinded outcome assessors will ensure unbiased data collection.

This study addresses the need for culturally responsive mental health interventions within Muslim populations. Ethical approval was obtained from the İstanbul Nişantaşı University Ethics Committee (Approval No: 20250103-27). Results are expected to contribute to evidence-based development of spiritually integrated psychotherapeutic models for anxiety and depression.

ELIGIBILITY:
Inclusion Criteria:

* Muslim individuals aged 18-65 years.
* Mild to moderate anxiety and/or depression symptoms (assessed via Beck
* Depression Inventory-II (BDI-II) and Beck Anxiety Inventory (BAI)).
* No formal psychiatric diagnosis but experiencing psychological distress.
* High religious belief levels, assessed via OK-Religious Attitude Scale.
* Not currently receiving psychotherapy or psychotropic medication.
* Ability to give informed consent and complete the study requirements.

Exclusion Criteria:

* Severe psychiatric disorders (schizophrenia, bipolar disorder, severe MDD).
* Current use of psychotropic medication or undergoing psychotherapy.
* History of substance abuse or dependence.
* Diagnosed dissociative disorders (contraindications for hypnosis).
* Cognitive impairment affecting comprehension of intervention.
* Severe medical conditions that may interfere with participation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-06-25 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory-II (BDI-II) | Baseline, Week 12 (post-intervention), Week 16 (follow-up)
  The study evaluates the effectiveness of Islamic-Oriented Ericksonian Hypnotherapy (IEH) vs. Standard Ericksonian Hypnotherapy (SEH) vs. No Intervention in reducing depressive symptoms. Depression severity will be assessed using the Beck Depression Inventory-II (BDI-II), comparing baseline, post-intervention (Week 12), and follow-up (Week 16) scores.
Beck Anxiety Inventory (BAI) | Baseline, Week 12, Week 16
  The study measures reductions in anxiety symptoms among participants receiving IEH, SEH, or no intervention. Anxiety severity will be assessed using the Beck Anxiety Inventory (BAI), comparing scores from baseline to post-intervention and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Metin Çınaroğlu, Phd, Principal Investigator — Istanbul Nisantasi Universitesi
Locations (1):
- İstanbul Nişantaşı University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) will be shared upon publication of the study results in a peer-reviewed journal. The shared dataset will include anonymized scores from outcome measures (e.g., BDI-II, BAI) and will exclude any personally identifiable information. Data will be available upon reasonable request for research purposes.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD and supporting information will be available after publication of study results and will remain accessible for five years post-publication.
Access Criteria: Researchers requesting access must submit a formal request specifying their intended use of the data. Access will be granted upon institutional review and approval by the research team. Requests can be made by contacting the corresponding author via email.